CLINICAL TRIAL: NCT02863588
Title: Determination of Genetic Susceptibility in Severe Recurrences of Ocular Toxoplasmosis
Acronym: TREXO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6433
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Toxoplasmosis Infection; Genotype II; Ocular Toxoplasmosis With Recurrences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- seropositive for Toxoplasma gondii (Experimental)
  Interventions: Biological: seropositive for Toxoplasma gondii

INTERVENTIONS:
Biological: seropositive for Toxoplasma gondii — blood sample

SUMMARY:
Ocular toxoplasmosis (OT) is a major cause of visual impairment worldwide. OT is responsible for 30 to 50% of posterior uveitis. It is characterized by dormant infections that may reactivate without known reasons, causing severe irreversible visual loss. The overall recurrence rate of OT in Europe is greater than 80% for patients and may range from one episode to 11 episodes (1% of OT) in the most extreme cases. Current treatments do not reduce the risk of recurrences and the risk of toxoplasmosis recurrence cannot be predicted in these immunocompetent patients. These clinical and biological expression changes might be related to an individual genetic susceptibility of each patient. The advanced analysis of the entire genome now possible to consider the project.

ELIGIBILITY:
Inclusion Criteria:

* seropositive for Toxoplasma gondii (for patient and parents)
* Infection with genotype II (for patient and parents)
* ocular toxoplasmosis recurrences >5 (patients only)

Exclusion Criteria:

* Parents seronegative for T. gondii infection
* Infection with others genotypes than type II

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Highlighting of genetic mutations associated with the susceptibility to Toxoplasma gondii.severe eye recurrences. Mutation analysis will be done by exome sequencing of the subjects included in this study | This analysis will be performed on a blood sample taken in patients included in the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud SAUER, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No